CLINICAL TRIAL: NCT06530537
Title: The Efficacy and Safety of Cilostazol Compared to Aspirin in Acute Non-Cardioembolic Stroke Patients With Concurrent Cerebral Microbleeds: An Open-Label, Endpoint-Blinded, Randomized Non-Inferiority Clinical Trial
Brief Title: Cilostazol vs. Aspirin in Acute Non-cardioembolic Stroke With Cerebral mIcrobleeds
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024083
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Microbleeds; Stroke
MeSH Terms: conditions — Stroke | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol Group (Experimental): Cilostazol 100mg twice daily
  Interventions: Drug: Cilostazol
- Aspirin Group (Active Comparator): Aspirin 100mg once daily
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100mg twice daily
  Arms: Cilostazol Group
Drug: Aspirin — Aspirin 100mg once daily
  Arms: Aspirin Group

SUMMARY:
The purpose of this clinical trial is to demonstrate that cilostazol is non-inferior to aspirin in terms of efficacy and safety for the secondary prevention of stroke in patients with acute non-cardioembolic ischemic stroke who have concurrent microbleeds. Researchers will compare the medication cilostazol with aspirin to assess its efficacy and safety in these patients.

Participants will:

Take the medication cilostazol or aspirin daily as part of an antiplatelet drug therapy.

Have baseline data and follow-up data collected at the time of hospital admission, and then at 3 months, 6 months post-discharge, and annually thereafter up to 4 years.

Have the primary endpoint set as stroke recurrence, with secondary endpoints being composite vascular events. Safety events will include moderate to severe hemorrhage and bleeding at any site.

DETAILED DESCRIPTION:
The plan is to enroll patients with acute non-cardioembolic stroke who have concurrent cerebral microbleeds (CMBs). After enrollment, patients will be randomly assigned to either the Cilostazol group (experimental group, Cilostazol 100mg, twice daily) or the Aspirin group (control group, Aspirin 100mg, once daily). The treatment goals for blood pressure, blood sugar, and blood lipids will be strictly controlled according to the relevant guidelines. Baseline and follow-up data will be collected at the time of enrollment, and at 3 months, 6 months, and annually (up to 4 years) after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke (within 1 month of onset)
* Non-cardioembolic stroke
* Presence of cerebral microbleeds (CMBs) confirmed by susceptibility-weighted imaging (SWI)

Exclusion Criteria:

* Previous diagnosis of cerebral amyloid angiopathy (CAA) according to the Boston 2.0 diagnostic criteria
* History of intracerebral hemorrhage highly suspected to be caused by CAA-related lobar hemorrhage
* Severe adverse reactions (such as active bleeding, severe allergies, etc.) to aspirin or cilostazol in the past, leading to non-compliance with medication
* Requirement for combined anticoagulant therapy
* Requirement for long-term dual antiplatelet therapy (>1 month)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2031-08-30 (Estimated); Study Completion 2031-08-30 (Estimated)

PRIMARY OUTCOMES:
The rate of recurrent stroke | Time Frame: baseline ,3-month,6-month, and every 1 year, follow-up time up to 4 years
  Head CT,Brain MRI,Cognitive Evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No